CLINICAL TRIAL: NCT01915849
Title: A Randomized, Double-blinded, Placebo-controlled, Crossover Trial to Assess the Effect of Orally Administered LIK066 on Glucose Absorption in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of LIK066 on Glucose Absorption in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: CLIK066A2201
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Results first posted 2015-02-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — licogliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1: LIK066 15 mg/Placebo/LIK066 50 mg/LIK066 150 mg (Experimental): Period 1- LIK066 15 mg treatment once daily (q.d.) for 4 days. Period 2- Placebo treatment once daily for 4 days Period 3 - LIK066 50 mg treatment once daily (q.d.) for 4 days. Period 4- LIK066 150 mg treatment once daily (q.d.) for 4 days. 14 days washout periods between treatment periods.
  Interventions: Drug: LIK066; Drug: Placebo
- Sequence 2: LIK066 50 mg/LIK066 15 mg/LIK066 150 mg/Placebo (Experimental): Period 1- LIK066 50 mg treatment once daily (q.d.) for 4 days. Period 2- LIK066 15 mg treatment once daily (q.d.) for 4 days. Period 3- LIK066 150 mg treatment once daily (q.d.) for 4 days. Period 4- Placebo treatment once daily for 4 days. 14 days washout periods between treatment periods.
  Interventions: Drug: LIK066; Drug: Placebo
- Sequence 3: LIK066 150 mg/LIK066 50 mg/Placebo/LIK066 15 mg (Experimental): Period 1- LIK066 150 mg treatment once daily (q.d.) for 4 days. Period 2- LIK066 50 mg treatment once daily (q.d.) for 4 days. Period 3- Placebo treatment once daily for 4 days. Period 4- LIK066 15 mg treatment once daily (q.d.) for 4 days. 14 days washout periods between treatment periods.
  Interventions: Drug: LIK066; Drug: Placebo
- Sequence 3: Placebo/LIK066 150 mg/LIK066 15 mg/LIK066 50 mg (Experimental): Period 1- Placebo treatment once daily (q.d.) for 4 days. Period 2- LIK066 150 mg treatment once daily (q.d.) for 4 days. Period 3- LIK066 15 mg treatment once daily (q.d.) for 4 days. Period 4- LIK066 50 mg treatment once daily (q.d.) for 4 days. 14 days washout periods between treatment periods.
  Interventions: Drug: LIK066; Drug: Placebo

INTERVENTIONS:
Drug: LIK066 — LIK066 15 mg, 50 mg and 150 mg
Drug: Placebo

SUMMARY:
The purpose of the study was to assess the effect of LIK066 on intestinal glucose absorption immediately after a single dose (immediate effect) and 6 hours following the dose (after multiple daily doses; sustained effect) in patients with type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Patients, age 18-65 years, must have been diagnosed with T2DM at least 6 months prior to screening with HbA1c 6.5 to 10.0%, inclusive, at screening.
* Fasting plasma glucose ≤250mg/dL at screening.
* If treated with metformin, patients must be on a stable dose for 12 weeks prior to randomization and maintain the dose until the end of the study.

Exclusion Criteria:

* Patients with type 1 diabetes mellitus.
* Patients with history of acute diabetic complications within the 6 months prior to screening.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential unless they are using effective methods of contraception during dosing of study treatment.
* Patients with signs or symptoms of significant diabetic complications.
* Patients treated with certain blood pressure or lipid lowering medications unless patients have been on stable doses for the 12 weeks prior to dosing.
* History of drug or alcohol abuse within the 12 months prior to dosing.
* Any surgical or medical condition, acute or unstable chronic disease which may, based on the investigator's opinion, jeopardize the patient in case of participation in the study.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Chula Vista, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: LIK066 15 mg/Placebo/LIK066 50 mg/LIK066 150 mg: Period 1- LIK066 15 mg treatment once daily (q.d.) for 4 days. Period 2- Placebo treatment once daily for 4 days. Period 3 - LIK066 50 mg treatment once daily (q.d.) for 4 days. Period 4- LIK066 150 mg treatment once daily (q.d.) for 4 days. 14 days washout periods between treatment periods.
- Sequence 4: Placebo/LIK066 150 mg/LIK066 15 mg/LIK066 50 mg: Period 1- Placebo treatment once daily (q.d.) for 4 days. Period 2- LIK066 150 mg treatment once daily (q.d.) for 4 days. Period 3- LIK066 15 mg treatment once daily (q.d.) for 4 days. Period 4- LIK066 50 mg treatment once daily (q.d.) for 4 days. 14 days washout periods between treatment periods.
Period: Treatment Period 1 (4 Days)
Arm/Group | Sequence 1: LIK066 15 mg/Placebo/LIK066 50 mg/LIK066 150 mg | Sequence 2: LIK066 50 mg/LIK066 15 mg/LIK066 150 mg/Placebo | Sequence 3: LIK066 150 mg/LIK066 50 mg/Placebo/LIK066 15 mg | Sequence 4: Placebo/LIK066 150 mg/LIK066 15 mg/LIK066 50 mg
Started | 5 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Treatment Period 2 (4 Days)
Arm/Group | Sequence 1: LIK066 15 mg/Placebo/LIK066 50 mg/LIK066 150 mg | Sequence 2: LIK066 50 mg/LIK066 15 mg/LIK066 150 mg/Placebo | Sequence 3: LIK066 150 mg/LIK066 50 mg/Placebo/LIK066 15 mg | Sequence 4: Placebo/LIK066 150 mg/LIK066 15 mg/LIK066 50 mg
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 3 (4 Days)
Arm/Group | Sequence 1: LIK066 15 mg/Placebo/LIK066 50 mg/LIK066 150 mg | Sequence 2: LIK066 50 mg/LIK066 15 mg/LIK066 150 mg/Placebo | Sequence 3: LIK066 150 mg/LIK066 50 mg/Placebo/LIK066 15 mg | Sequence 4: Placebo/LIK066 150 mg/LIK066 15 mg/LIK066 50 mg
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4 (4 Days)
Arm/Group | Sequence 1: LIK066 15 mg/Placebo/LIK066 50 mg/LIK066 150 mg | Sequence 2: LIK066 50 mg/LIK066 15 mg/LIK066 150 mg/Placebo | Sequence 3: LIK066 150 mg/LIK066 50 mg/Placebo/LIK066 15 mg | Sequence 4: Placebo/LIK066 150 mg/LIK066 15 mg/LIK066 50 mg
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: all patients that received study drug and with no protocol deviations with relevant impact on safety.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: LIK066 15 mg/Placebo/LIK066 50 mg/LIK066 150 mg | Sequence 2: LIK066 50 mg/LIK066 15 mg/LIK066 150 mg/Placebo | Sequence 3: LIK066 150 mg/LIK066 50 mg/Placebo/LIK066 15 mg | Sequence 4: Placebo/LIK066 150 mg/LIK066 15 mg/LIK066 50 mg | Total
Number analyzed (Participants) | 5 | 3 | 3 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.4 (9.29) | 54.0 (10.54) | 62.3 (3.06) | 56.0 (8.19) | 56.0 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 1 | 7
  Male | 2 | 2 | 1 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Postprandial Curve (AUC) for Rate of Appearance (Ra) of Exogenous Glucose
Description: Glucose fluxes during a mixed meal were measured using a dual glucose tracer method and non-steady state Steele equations. The rate of appearance of meal (or exogenous) glucose in the blood (also referred to as intestinal glucose absorption or Ra meal) after a mixed meal following LIK066 administration on Days 1 and 4 was the primary PD assessment in this study.The postprandial AUC was calculated using the linear trapezoidal rule. The sample collected at 7 hours after the start of the infusion was treated as the pre-meal, 0 hour measurement for the AUC0-5 hr calculation.
Time Frame: Day 1 and Day 4 (pre-meal, every half hour till 5 hour on Day 1 and Day 4)
Population: The pharmacodynamic (PD) analysis set included all patients with any available PD data, who received any study drug and experienced no protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: (umol/kg FFM/min)*hr
Groups:
- LIK066 15 mg: All patients who have received LIK066 15 mg once daily for 4 days.
- LIK066 50 mg: All patients who have received LIK066 50 mg once daily for 4 days.
- LIK066 150 mg: All patients who have received LIK066 150 mg once daily for 4 days.
- Placebo: All patients who have received placebo once daily for 4 days.
Arm/Group | LIK066 15 mg | LIK066 50 mg | LIK066 150 mg | Placebo
Number analyzed (Participants) | 14 | 12 | 12 | 11
(umol/kg FFM/min)*hr
  Day 1 | 101.97 (29.348) | 93.89 (25.852) | 63.84 (22.589) | 97.76 (30.615)
  Day 4 | 109.99 (27.144) | 117.81 (30.881) | 112.45 (31.129) | 103.97 (23.335)

ADVERSE EVENTS:
Description: Safety analysis set: all patients that received study drug and with no protocol deviations with relevant impact on safety.
Groups:
- Placebo: Placebo
- LIK066 15 mg: LIK066 15 mg
- LIK066 50 mg: LIK066 50 mg
- LIK066 150 mg: LIK066 150 mg
Arm/Group | Placebo | LIK066 15 mg | LIK066 50 mg | LIK066 150 mg
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 8/14 | 7/12 | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | LIK066 15 mg (N=14) | LIK066 50 mg (N=12) | LIK066 150 mg (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 8
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 4
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Cyst (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Implant site haemorrhage (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Vulvovaginitis (Infections and infestations) | 0 | 0 | 1 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.